CLINICAL TRIAL: NCT01640886
Title: Prospective Study Into the Performance of the KeyPathtm MRSA/MSSA Blood Culture Test - BTA
Brief Title: Study of the Performance of the KeyPath MRSA/MSSA Blood Culture Test - BTA
Status: Terminated | Type: Observational
Why Stopped: Results did not meet study requirements.
Sponsor: MicroPhage, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MP2012-A
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Bacteremia
Keywords: Staphylococcus aureus; methicillin resistant; MRSA; MSSA; Blood Culture; Diagnostic
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retention of de-identified blood culture specimens only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of Care: 1. Comparison of S. aureus to the reference methods for S. aureus (tube coagulase and Staphaurex.)
  2. Comparison to the reference method (30 ug cefoxitin disc diffusion).
- KeyPath Test Group: All specimens collected that meet the inclusion criteria will be tested using the KeyPath BTA Test.

SUMMARY:
In vitro identification of S. aureus,methicillin-sensitive S. aureus (MSSA) and methicillin-resistant S. aureus (MRSA)from positive blood culture using MicroPhage's bacteriophage-based diagnostic platform.

DETAILED DESCRIPTION:
This is a multi-center clinical study to investigate the effectiveness of the performance of the KeyPath MRSA/MSSA Blood Culture Test - BTA. The KeyPath test is performed directly on positive blood culture specimens from bioMerieux BacT/ALERT blood culture bottles. The MicroPhage test will be compared to standards and market available tests with similar indications (comparators). It is estimated that the study will last 3-4 months depending on the accural rate at the institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Blood culture samples determined to be Gram-positive from subjects aged 18+, inclusive, with any of the following bottle types:

   * bioMerieux BacT/ALERT® Standard Aerobic and Anaerobic
   * bioMerieux BacT/ALERT® FAN Aerobic and FAN Anaerobic
2. Completion of the KeyPathTM BTA Test on the sample.
3. Completion of the reference method for S. aureus identification (tube coagulase and Remel Staphaurex ) and completion of the reference method for methicillin resistance determination (30 µg cefoxitin disc diffusion) for S. aureus positive samples.

Exclusion Criteria:

1. Samples from blood culture positives over 24 hours from alarm
2. Samples deemed contaminated.
3. Violations and/or deviations from the KeyPathTM BTA Test protocol and/or other included test protocols under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients with Gram positive blood cultures determined to be positive with the following bottle types:
  1. bioMerieux BacT/Alert Standard Aerobic and Anaerobic
  2. bioMerieux BacT/Alert FAN Aerobic and FAN Anaerobic
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prospective study into the performance of the KeyPath MRSA/MSSA Blood Culture Test -BTA | 3-4 months
  A. Determination of the performance of the KeyPathTM MRSA/MSSA Blood Culture Test - BTA for identification of S. aureus and determination of MRSA and MSSA direct from clinical blood culture positives by:
  i. KeyPathTM MRSA/MSSA Blood Culture Test - BTA for identification of S. aureus to the reference methods for S. aureus (tube coagulase and Staphaurex).
  ii. KeyPathTM MRSA/MSSA Blood Culture Test - BTA for determination of MRSA and MSSA among S. aureus positives by comparison to the reference method (30 µg cefoxitin disc diffusion).

CONTACTS AND LOCATIONS:
Overall Officials: Dipankar Manna, Ph.D., Principal Investigator — MicroPhage, Inc.
Locations (3):
- United States (3):
  - University of Arizona, Infectious Disease Research, Tuscon, Arizona
  - UCLA Clinical Laboratory, Los Angeles, California
  - Medical University of South Carolina, Charleston, South Carolina